CLINICAL TRIAL: NCT00574353
Title: A Feasibility Study Using Fluorine-18-Labeled Fluoro-Misonidazole Positron Emission Tomography to Detect Hypoxia in Locally Advanced (T3-T4 and./or N1)Primary Rectal Cancer Patients
Brief Title: Study Using Fluorine-18-Labeled Fluoro-Misonidazole Positron Emission Tomography to Detect Hypoxia in Locally Advanced (T3-T4 and./or N1)Primary Rectal Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 07-151
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; 07-151
MeSH Terms: conditions — Colorectal Neoplasms

ARMS (1):
- 1 (Experimental): FMISO PET study.
  Interventions: Radiation: Fluorine-18-Labeled Fluoro-Misonidazole Positron Emission

INTERVENTIONS:
Radiation: Fluorine-18-Labeled Fluoro-Misonidazole Positron Emission — You will be scanned 2 to 3 times on the same day, but you will only be administered one dose of the FMISO tracer. The first scan will last about 30 minutes. Then you will have 1 to 3 hours to wait before you are scanned again. Some patients will undergo a second scan approximately one-and-a-half hours after the start of the first scan. This scan will last about 10 minutes. The final scan will occur between 2-4 hours after the start of the first scan. This final scan will also last about 10 minutes. During the PET scan, you may have a separate i.v. line put into your other arm so that we can take 2 to 3 blood samples. These samples will be less than half a teaspoon each. We are taking these blood samples to see how quickly FMISO leaves your blood stream. The first sample will be taken between 2 and 40 minutes after the FMISO is injected. The other two blood samples will be taken with each subsequent scan.

SUMMARY:
When used with a different radioactive tracer called FMISO, a PET scan can find areas of low oxygen in the tumor. We think that having areas of low oxygen is a reason why some tumors are hard to treat with radiation.

In a past study, FMISO PET scans were performed in 6 patients with rectal cancer that could not be operated on and that had spread to other areas. In this group of patients, FMISO PET scans were able to find the low oxygen areas in their tumors. But this study included only a few patients. In the present study, we want to use FMISO PET scans in patients who have tumors that can be operated on. This group of patients will have radiation, chemotherapy or both before they have their surgery. We want to see if FMISO PET can find low oxygen areas in this distinct group of patients.

DETAILED DESCRIPTION:
Hypoxia is a characteristic feature of malignant solid tumors associated with poor prognosis and resistance to chemotherapy and radiation. It has also been shown (6) that the presence of hypoxia may reduce long-term survival post surgery. Hypoxia renders tumor cells up to three times more resistant to ionizing radiation than aerobic cells. The presence of hypoxic regions within tumors may be one factor leading to local failure after treatment with standard pre-operative radiotherapy doses. If these regions could be identified and verified using a non-invasive imaging technique prior to surgery, they could be specifically targeted using sophisticated planning techniques such as intensity modulated radiation therapy (IMRT) to deliver higher doses ionizing radiation with preoperative radiotherapy. Future studies using IMRT to "dose paint" areas of hypoxia within tumors will build upon the results of this feasibility study. Ultimately, by the delivery of differential dose of radiation to the tumor, in combination with surgery, the local control rates of rectal cancer patients may further be improved.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Histologically confirmed diagnosis of Stage 2 or Stage 3 rectal carcinoma requiring preoperative radiation, chemotherapy or both, per treating physician
* 18 years of age or older
* Karnofsky performance status ≥ or = to 70

Exclusion Criteria:

* Women who are pregnant (confirmed by serum b-HCG in women of reproductive age) or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-12-11 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Humm, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- FMISO PET Study: FMISO PET study.
  Fluorine-18-Labeled Fluoro-Misonidazole Positron Emission
Period: Overall Study
Arm/Group | FMISO PET Study
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FMISO PET Study
Number analyzed (Participants) | 23
Age, Continuous [Mean (Full Range); unit: years] | 54 [35 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 19
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Successfully Scanned Using F-FMISO-PET Imaging
Description: The uptake kinetics of [18F]-Fluoromisonidazole activity in the colorectal lesion was entered into a compartmental model to determine the rate constants of uptake (k1) and irreversible binding (k3) in the lesion on the PET scan at different times post injection. Also the tumor to background ratio was determine. A plot of k3 and TNB was plotted. This will help determine the Feasibility of a Non-invasive Method of Detecting Hypoxia, Using F-FMISO-PET Imaging in Colorectal Cancer Patients.
Time Frame: Post injection between 0-30 min, and again at the nominal times of 90 min and 180 min
Measure: Count of Participants; unit: Participants
Arm/Group | FMISO PET Study
Number analyzed (Participants) | 23
Participants
  Participants successfully scanned | 18
  Participants not scanned | 5

2. Secondary Outcome: Number of Participants Who Had Blood Samples Collected
Description: Blood sample was taken in order to determine the blood pharmacokinetics of [18F]-Fluoromisonidazole in these participants.
Time Frame: Up to 180 minutes post injection
Measure: Count of Participants; unit: Participants
Arm/Group | FMISO PET Study
Number analyzed (Participants) | 23
Participants
  Blood sample collected | 10
  Blood sample was not collected | 13

ADVERSE EVENTS:
Time Frame: 180 minutes post injection
Arm/Group | FMISO PET Study
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT00574353/Prot_SAP_000.pdf